CLINICAL TRIAL: NCT07182786
Title: The Efficacy of Laryngeal Mask Airway Gastro (LMA® Gastro™) in Preventing Hypercarbia in ERCP Patients: A Randomized Controlled Study
Brief Title: The Efficacy of Laryngeal Mask Airway Gastro (LMA® Gastro™) in Preventing Hypercarbia in ERCP Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Karim Mohamed Aly Ahmed, Assistant Lecturer of Anesthesiology, Surgical ICU & Pain Management,Theodor Bilharz Research Institute. Candidate for MD degree , Anaesthesia department , Cairo University., Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MD-507-2023
Record Dates: First submitted 2025-09-05; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Endoscopy, Gastrointestinal; Procedural Sedation; Anesthesia Airway Management; Anesthesia for Endoscopic Procedures
Keywords: ERCP anesthesia; Anesthesia for endoscopy; LMA Gastro; Hypercarbia
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LMA Gastro group (L group): total intravenous anesthesia and LMA Gastro (Active Comparator)
  Interventions: Device: LMA Gastro
- Control group (C group): total intravenous anesthesia with no airway device , with Nasal Cannula. (No Intervention)

INTERVENTIONS:
Device: LMA Gastro — LMA Gastro, is a laryngeal mask airway device that is specifically designed for air way management in GIT endoscopic procedures due to having a channel dedicated for endoscope introduction. the safety and efficacy of LMA Gastro was researched in many studies, but its role in preventing Hypercarbia during ERCP procedures is yet to be researched and tested.
  Arms: LMA Gastro group (L group): total intravenous anesthesia and LMA Gastro

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) has evolved into a primarily therapeutic procedure that often requires anesthetic support. While moderate to deep sedation is commonly used, it carries a high risk of respiratory complications, including hypoxemia and hypercapnia, which can lead to cardiovascular instability. General anesthesia with endotracheal intubation offers greater airway protection but is associated with hemodynamic stress, the need for neuromuscular blockade, longer recovery, and potential airway trauma.

The LMA® Gastro™ Airway, introduced in 2017, was specifically designed for upper gastrointestinal endoscopy. It combines a supraglottic airway with a dedicated channel for the endoscope, enabling ventilation and airway protection while facilitating the procedure. Early studies demonstrate high success rates for both airway management and ERCP completion, with a low incidence of adverse events. However, most available evidence is observational, and randomized controlled trials are needed to establish its effectiveness compared with traditional sedation and general anesthesia with intubation.

In conclusion, the LMA Gastro shows promise as a safe and efficient alternative airway device for ERCP, potentially bridging the gap between deep sedation and invasive intubation, though further evidence is required to confirm its impact on respiratory and hemodynamic outcomes.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) is fast emerging as a therapeutic procedure rather than a diagnostic one, requiring anesthetic support for successful completion of the procedure. The procedure can be uncomfortable especially due to prone positioning, multiple passages of endoscope, air insufflations, dilatation of ductal structures and prolonged duration which requires a high degree of cooperation from patients. A large number of patients need to be given general anesthesia (GA), in order to minimize incidence of adverse respiratory and hemodynamic events in the peri-procedure period. The use of GA with endotracheal intubation (ETT) or supraglottic devices protects the airway, reduces ERCP failure and complication rates. However, ETT involves rigid laryngoscopy with consequent undesirable hemodynamic responses and use of neuromuscular blocking drugs. It also has the disadvantage of a longer recovery time and possibility of injury to the oro-pharynx at insertion.

Moderate to deep sedation is a commonly employed technique for ERCPs, with general anesthesia utilizing an endotracheal intubation being reserved for selected cases. Reported rates of hypoxemia during all endoscopic procedures range from 11 to 50%, and this may be as high as 60% with ERCP. Sustained hypoxia is a major risk factor for peri-procedural cardiac arrhythmias and myocardial ischemia. Respiratory complications that occur during intravenous sedation have a higher risk of hypercapnia than hypoxemia. Patients receiving propofol-based tubeless sedation may be at higher risk of sedation-related adverse events than patients receiving GA. Moreover, when low-flow oxygen is administered through a nasal cannula, the apparent oxygen saturation value is maintained at a normal concentration; however, hypoventilation is sustained, which may result in impaired exhalation. Gradual CO₂ accumulation, and CO₂ concentrations maintained at 60 mmHg or higher, are risk factors for secondary circulatory abnormalities such as an abnormal increase in blood pressure, tachycardia, and arrhythmia.

As the number of gastrointestinal endoscopic interventions and possibilities increased, and the number of patients with severe comorbidities and existing medical conditions, the need for minimally invasive airway devices specially dedicated for endoscopic procedures became relevant. A modified laryngeal tube with a dedicated channel for an endoscope was described as an alternative airway device. This approach was further developed with the introduction of the LMA® Gastro™ Airway, a refined tool in advanced airway management for upper gastrointestinal endoscopy.

The LMA® Gastro™ Airway is a cuffed peri-laryngeal supraglottic airway (SGA) with an endoscopic channel, having a maximum diameter of 14 mm, which suits all standard endoscopes. Its design features include a channel for esophageal intubation, a separate channel with a terminal cuff for lung ventilation, and an integrated bite block and cuff pressure indicator. It comes in three available sizes: #3 (30-50 kg), #4 (50-70 kg), and #5 (70-100 kg).

This device has been reported to have a high airway insertion success rate and a high first-attempt endoscopy success rate in patients with low risk of pulmonary aspiration. Observational studies have suggested that the LMA Gastro may be a safe alternative to tubeless anesthesia in patients undergoing ERCP, though some were limited by small sample size and non-randomized design. Retrospective analyses have demonstrated high success rates of ERCP completion with well-maintained ventilation and minimal intraoperative and postoperative adverse events. However, confounding factors in patient selection and the absence of randomized controlled comparisons with conventional airway techniques remain limitations.

Although the LMA Gastro has been demonstrated in several studies as a safe and efficient substitute for general anesthesia or deep sedation tubeless anesthesia for ERCP procedures, to date there is no exact measurement or assessment of its role in prevention of hypercarbia or hypoxia.

Aim of the work:

The aim of this study is to evaluate the efficacy of using LMA Gastro in preventing hypercarbia and decreasing hypoxic and hyper carbic episodes in patients undergoing ERCP procedures of average timing and difficulty according to the ASGE (American Society of Gastroenterologists) grading system. In addition, to assess the efficiency of using the new LMA Gastro® airway device in endoscopic procedures and its stress response.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age: 20-45 years
* ASA classification: II and III
* Body mass index: 25 -30 kg/m2
* Height > 155 cm
* ERCP procedures of difficulty grade II and III (according to American Society of Gastroenterologists ASGE grading system for ERCP procedures).

Exclusion Criteria:

* Anticipated difficult airway
* Restricted head and neck mobility
* Pulmonary disease
* Obese Patients with a BMI of ≥ 35 kg/m2
* Patients with moderate to severe ascites
* Patients with Childe-Pughe-Turcotte (CPT) classification C
* Increased risk of aspiration (for example incomplete fasting hours, delayed gastric emptying, gastric outlet obstruction, etc.)
* ERCP procedures of difficulty grade I (due to relatively short procedure duration)
* ERCP procedures of malignant obstructive jaundice
* ERCP procedures less than 30 minutes and more than 120 minutes.
* Patient refusal

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
End tidal CO2 | 30 minutes from induction of Anesthesia
  End tidal CO2 measurement after 30 minutes of procedure time. It is measured by capnography in patients undergoing ERCP procedure.

SECONDARY OUTCOMES:
Hypercarbia | Procedures of duration between 30 and 120 minutes
  ETCO2 (≥45 mmHg) or PaCO2(≥50 mmHg) or both Highest ETCO2 and PaCO2 recorded during procedure
Timing of Hypercarbia | Procedures of duration between 30 and 120 minutes
  Time till ETCO2 (≥45 mmHg) or PaCO2(≥50 mmHg) or both
Hypoxia | Procedures of duration between 30 and 120 minutes.
  Lowest SpO2 and PaO2 recorded during procedure
Number of Hypoxic episodes | Procedures of duration between 30 and 120 minutes
  Number of hypoxic episodes (desaturation to SPO2 of 92% or below for at least 15 seconds)
Hemodynamic stress response : Heart Rate | Procedures of duration between 30 and 120 minutes.
  Heart rate
Hemodynamic stress response : Mean arterial blood pressure | Procedures of duration between 30 and 120 minutes.
  Mean arterial blood pressure
Efficiency of LMA gastro in anesthesia of ERCP procedures: duration till endoscope introduction. | From Anesthesia induction till start of procedure
  Measuring time taken from induction of anesthesia till ERCP duodenoscope introduction( start of ERCP procedure).
Efficiency of LMA gastro in anesthesia of ERCP procedures: Ease of duodenoscope introduction. | From induction of Anesthesia till start of procedure
  Number of attempts of ERCP duodenoscope introduction
Efficiency of LMA gastro in anesthesia of ERCP procedures: ease of LMA Gastro insertion. | From induction of Anesthesia till start of procedure
  Number of attempts of LMA Gastro insertion
Efficiency of LMA gastro in anesthesia of ERCP procedures: Safety of LMA Gastro | During whole ERCP procedure
  Number of displacements of LMA Gastro and need for repositioning
Efficiency of LMA gastro in anesthesia of ERCP procedures: Anesthetic consumption of propofol | whole duration of ERCP procedure
  * Mean dose of propofol used in induction in both groups
  * Mean dose of propofol used for maintenance of anesthesia
Efficiency of LMA gastro in anesthesia of ERCP procedures: Recovery time | from the end of ERCP procedure till discharge to PACU
  Recovery time (from stopping propofol infusion till discharge to PACU)
Efficiency of LMA gastro in anesthesia of ERCP procedures: procedure failure | procedures between 30 and 120 minutes
  Number of failed procedures in both groups
Efficiency of LMA gastro in anesthesia of ERCP procedures: procedure duration | procedures between 30 and 120 minutes
  Effect of using LMA Gastro on average procedure duration in comparison to control group
Efficiency of LMA gastro in anesthesia of ERCP procedures: post operative complications | From end of procedure till discharge from PACU (after 30 min.)
  occurrence of post operative Nausea, vomiting or sore throat
Efficiency of LMA gastro in anesthesia of ERCP procedures: operator satisfaction | procedures between 30 and 120 minutes
  The operator rates the following on a scale from 1to 5 ( 1 being worst and 5 the best):
  * ease of endoscope introduction
  * ease of manipulation and advancement
  * overall satisfaction
Efficiency of LMA gastro in anesthesia of ERCP procedures: anesthesiologist satisfaction | procedures between 30 and 120 minutes
  The anesthesiologist rates the following on a scale from 1 to 5 ( 1 being the worst and 5 the best):
  * ease of LMA Gastro insertion
  * overall satisfaction
Efficiency of LMA gastro in anesthesia of ERCP procedures: conversion to endotracheal intubation. | procedures between 30 and 120 minutes
  number of procedures that were converted to traditional endotracheal intubation due to vomiting, risk of aspiration with excessive secretions in oral cavity, severe laryngeal spasm not responding to increasing depth of anesthesia or I.V. lidocaine, airway obstruction and persistent hypoxia.

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided